CLINICAL TRIAL: NCT03693638
Title: A Comparative Study of Fractionated Vs Single Dose Injection for Spinal Anesthesia During Caesarean Section in Patients With Pregnancy-Induced Hypertension
Brief Title: Fractionated Vs Single Dose Injection for Spinal C-Section in Patients With Pregnancy-Induced Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Alfan Mahdi Nugroho, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes024
Record Dates: First submitted 2018-09-26; First posted 2018-10-03 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy Induced Hypertension
Keywords: spinal anesthesia; pregnancy-induced hypertension; Cesarean section
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single dose (SD) (Active Comparator): 2,5 ml total anesthetic drug dose (Bupivacaine-fentanyl) were given with 0.2 ml/second rate, and subjects were asked to remain sitted for 90 seconds
  Interventions: Drug: Bupivacaine-fentanyl
- Fractionated dose (FD) (Active Comparator): 1,5 ml of total anesthetic drug dose (Bupivacaine-fentanyl) followed by 1 ml remaining dose after 90 s interval were given
  Interventions: Drug: Bupivacaine-fentanyl

INTERVENTIONS:
Drug: Bupivacaine-fentanyl — 2,5 ml total anesthetic drug dose were given with 0.2 ml/second rate, and subjects were asked to remain sitted for 90 seconds
  Arms: Single dose (SD)
Drug: Bupivacaine-fentanyl — 1,5 ml of total anesthetic drug dose followed by 1 ml remaining dose after 90 s interval were given
  Arms: Fractionated dose (FD)

SUMMARY:
The aim of this study was to compare haemodynamic changes, total dose of ephedrin requirement, and level of sensory blockade between fractionated dose and single dose spinal anesthesia injection in obstetric patients with pregnancy-induced hypertension who underwent Caesarean section

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study and randomized into two groups; single dose (SD) and fractionated dose (FD). All subjects will receive spinal anesthesia with 2,5 ml of 10 mg bupivacaine hyperbaric 0,5% and fentanyl 25 mcg. After IV cannulas (18 - 20 G) were properly placed, premedication with intravenous (IV) ranitidine 50 mg and metoclopramide 10 mg were given. Additional IV access was added if MgSO4 must been continuously administered intravenously perioperatively. Standard monitor device were placed after patients had been transferred to operating room. Additional premedication such as intravenous midazolam 0.02 mg/BW or fentanyl 1 mcg/BW were given if the patients were anxious or in pain. Baseline haemodynamic measurement was done two minutes after premedication. Spinal anesthesia was performed while patients in sitting position at L3-4 or L4-5 level with median or paramedian approach, with total dose 2,5 ml of 10 mg bupivacaine hyperbaric 0,5% and fentanyl 25 mcg. After skin wheal of lidocaine at the intended spinous interspace were placed, spinal needle (SpinocanR, B Braun, 27 G) were inserted and advanced until subarachnoid space were reached. In group FD, 1,5 ml of total dose followed by 1 ml remaining dose after 90 s interval were given. In SD group, 2,5 ml total dose were given with 0.2 ml/second rate, and subjects were asked to remain sitted for 90 seconds. If there were more than three injection attempts, the patients were excluded from the study. Co-loading 5 - 10 ml/kg ringer lactate in 20 minutes were given for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* with hypertension in pregnancy (gestational hypertension or preeclampsia)
* ASA II-III
* aged 18 - 40 years
* BMI 18.5 - 35 kg/m2
* singleton pregnancy
* would undergo spinal anesthesia for emergency or semi-emergency caesarean section

Exclusion Criteria:

* chronic hypertension
* eclampsia
* pulmonary edema
* cerebrovascular diseases
* type-2 diabetes mellitus and gestational diabetes
* placental abruption/previa/accreta
* umbilical cord prolapse
* gestational age <34 weeks
* estimated fetal weight <=2.300 gram and >=4.000 gram
* polyhydramnios
* fetal distress

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 42 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Change of mean arterial pressure (MAP) | 15 minutes
  drop of blood pressure more than 20% of baseline value, and were treated with ephedrine 5 - 10 mg which could be repeated if necessary

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chumpathong S, Chinachoti T, Visalyaputra S, Himmunngan T. Incidence and risk factors of hypotension during spinal anesthesia for cesarean section at Siriraj Hospital. J Med Assoc Thai. 2006 Aug;89(8):1127-32. PMID 17048420
- [Background] Sharwood-Smith G, Drummond GB. Hypotension in obstetric spinal anaesthesia: a lesson from pre-eclampsia. Br J Anaesth. 2009 Mar;102(3):291-4. doi: 10.1093/bja/aep003. No abstract available. PMID 19218369
- [Background] Badheka JP, Oza VP, Vyas A, Baria D, Nehra P, Babu T. Comparison of fractionated dose versus bolus dose injection in spinal anaesthesia for patients undergoing elective caesarean section: A randomised, double-blind study. Indian J Anaesth. 2017 Jan;61(1):55-60. doi: 10.4103/0019-5049.198390. PMID 28216705
- [Background] Hocking G, Wildsmith JA. Intrathecal drug spread. Br J Anaesth. 2004 Oct;93(4):568-78. doi: 10.1093/bja/aeh204. Epub 2004 Jun 25. No abstract available. PMID 15220175
- [Derived] Nugroho AM, Sugiarto A, Chandra S, Lembahmanah L, Septica RI, Yuneva A. A Comparative Study of Fractionated Versus Single Dose Injection for Spinal Anesthesia During Cesarean Section in Patients with Pregnancy-Induced Hypertension. Anesth Pain Med. 2019 Feb 6;9(1):e85115. doi: 10.5812/aapm-85115. eCollection 2019 Feb. PMID 30881909